CLINICAL TRIAL: NCT04980157
Title: CARES-HCV: Promoting Concurrent Hepatitis C Virus Screening and Colorectal Cancer Screening Uptake Among Diverse Baby Boomers
Brief Title: CARES-HCV: Promoting Screening Uptake Among Diverse Baby Boomers
Status: Completed | Type: Observational
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-20601
Record Dates: First submitted 2021-07-19; First posted 2021-07-28 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Hepatitis C Virus Infection; Colorectal Cancer
Keywords: HCV Screening; CRC Screening
MeSH Terms: conditions — Hepatitis C; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Patients born between 1945-1965 who have clinic visits at a partnering federally qualified health center.
  Interventions: Behavioral: CARES-HCV

INTERVENTIONS:
Behavioral: CARES-HCV — CARES-HCV is an educational intervention to promote both hepatitis c screening and colorectal cancer screening among diverse baby boomers in the area.

SUMMARY:
The purpose of the study is to examine the efficacy of educational materials to promote hepatitis C virus (HCV) screening and colorectal cancer (CRC) screening uptake among adults born between 1945-1965.

ELIGIBILITY:
Inclusion Criteria:

* Born between 1945 and 1965 and up to age 75
* No personal history of colorectal cancer (CRC) or current presumptive colorectal cancer symptoms (e.g., unresolved rectal bleeding or abdominal pain/bloating)
* No personal history of hepatitis C virus (HCV) or liver cancer
* Able to read, write, speak, and understand English or Spanish
* Not currently enrolled in another CRC screening or a HCV screening study
* At average risk for CRC (that is, no hereditary CRC syndromes such as lower gastrointestinal (GI) bleeding, persistent diarrhea, bloating, or lower GI pain, no strong family history of CRC)
* Not currently up-to date with CRC screenings
* Not having previously completed HCV screening
* Able and willing to complete a phone interview
* Able to provide informed consent

Ages: 56 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients born between 1945-1965 up to age 75 who have clinic visits at a partnering federally qualified health center.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Hepatitis C Virus (HCV) knowledge | Day 1 & Day 7
  Participants will be interviewed regarding their HCV knowledge on Day 1 prior to receiving educational materials. They will be interviewed once again approximately one week after receiving educational materials.
Change in Colorectal Cancer (CRC) knowledge | Day 1 & Day 7
  Participants will be interviewed regarding their CRC knowledge on Day 1 prior to receiving educational materials. They will be interviewed once again approximately one week after receiving educational materials.
Hepatitis C Virus Screening Status | at 6 months
  Data about participants' HCV screening status will be collected from Federally Qualified Health Care Center's (FQHC) 6 months after participants have received educational materials.
Colorectal Cancer Screening Status | at 6 months
  Data about participants' CRC screening status will be collected from Federally Qualified Health Care Center's (FQHC) 6 months after participants have received educational materials.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Christy, PhD, Principal Investigator — Moffitt Cancer Center; Clement K Gwede, PhD, MPH, RN, FAAN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided